CLINICAL TRIAL: NCT03622463
Title: A Randomized, Double-Blind, Placebo-controlled Trial of Antroquinonol in Patients With Atopic Dermatitis
Brief Title: A Trial of Antroquinonol in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHADERM-2-001
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Atopic Dermatitis
Keywords: Antroquinonol; Hocena
MeSH Terms: conditions — Dermatitis, Atopic | interventions — antroquinonol

STUDY DESIGN:
Intervention Model Description: This is a multi-centers, phase IIa, double blind, randomized, placebo-controlled trial of Antroquinonol in patients with atopic dermatitis. Subjects with diagnosis of atopic dermatitis, using the Hanifin and Rajka Diagnostic Criteria, who meet inclusion/exclusion criteria will be randomized into 3 groups:
  1. Antroquinonol 100 mg PO QD
  2. Antroquinonol 50 mg PO QD
  3. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antroquinonol 100 mg PO QD (Experimental): Antroquinonol (Hocena) 50mg/capsule. 2 capsules antroquinonol,once a day.
  Interventions: Drug: Antroquinonol
- Antroquinonol 50 mg PO QD (Experimental): Antroquinonol (Hocena) 50mg/capsule. 1 capsules antroquinonol and 1 capsule placebo, once a day.
  Interventions: Drug: Antroquinonol; Other: Placebo
- Placebo (Placebo Comparator): Placebo capsule, 2 capsules placebo, once a day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antroquinonol — Antroquinonol will be provided as a capsule-shaped which contain 50 mg Antroquinonol.
  Other Names: Hocena
  Arms: Antroquinonol 100 mg PO QD; Antroquinonol 50 mg PO QD
Other: Placebo — The matching placebo will be packaged as Antroquinonol with appearance identical in all aspects
  Arms: Antroquinonol 50 mg PO QD; Placebo

SUMMARY:
This is a multi-centers, phase IIa, double blind, randomized, placebo-controlled trial of Antroquinonol in patients with atopic dermatitis.Duration of treatment is 12 week in total. Study visits will occur every 4 weeks. AEs/SAEs, changes to concomitant medications will be noted, vital signs will be taken, and efficacy evaluations will be performed as well. The last estimation of variable scores will occur for all subjects.

DETAILED DESCRIPTION:
This is a multi-centers, phase IIa, double blind, randomized, placebo-controlled trial of Antroquinonol in patients with atopic dermatitis.Duration of treatment is 12 week in total. Study visits will occur every 4 weeks. During these visits study drug will be administered at the site, new AEs/SAEs as well as follow-up for AEs and SAEs that have not been resolved will be recorded, changes to concomitant medications will be noted, vital signs will be taken, and efficacy evaluations will be performed as well. The study includes collection of cytokines samples. The end-of-treatment visit and the last estimation of variable scores will occur at week 13 (visit 5) for all subjects. The final visit will be at week 15 (visit 6). Subjects will be encouraged to complete all planned visits regardless of their adherence to study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 20 and 65 years who had moderate-to-severe atopic dermatitis (using the Hanifin and Rajka Diagnostic Criteria)
* Patients with body weight ≥ 25 kg and ≤ 120 kg, singing informed consent
* To be eligible to participate, patients were required to havea.

  1. score of at least 5 on the Eczema Area and Severity Index (EASI), which rangesfrom 0 to 72, with higher scores indicating worse disease severity;
  2. a score for pruritus of at least 30 mm on a visual-analogue scale, which ranges from 0 (no itch) to 100 mm (worst itch imaginable);
  3. a score of at least 2 on the static Investigator's Global Assessment (sIGA), which ranges from 0 (clear) to 4 ( severe disease).
  4. BSA affected or PSAI ≥ 5%

Exclusion Criteria:

1. Patients with active dermatologic diseases concomitant with atopic dermatitis.
2. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
3. Subjects with defective epidermal barrier(e.g Netherton's syndrome)
4. Any subject who is immunocompromised or has a history of malignant disease. This information will be gathered verbally from the patient while taking a medical history from the patient, and will not involve further testing such as an HIV test.
5. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
6. Any noticeable breaks or cracks in the skin on either arm, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
7. Ongoing participation in another investigational trial
8. Use of any oral or topical antibiotic for up to four weeks prior to the reatment visit or active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
9. Use of any systemic immunosuppressive therapy (e.g. CsA, MTX, etc.) within four weeks of the Treatment visit.
10. Participant who has a condition or is in a situation that, in the investigator's opinion, may put the patient at significant risk, or may significantly interfere with the patient's participation in the study.
11. Subjects with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices.
12. History of food or drug related severe anaphylactoid or anaphylactic reaction(s)
13. Pregnancy or breast feeding
14. History or presence of epilepsy, significant neurological disorders, cerebrovascular attack or ischemia
15. History or presence of myocardial infarction or cardiac arrhythmia under drug therapy
16. Patients who are unable to complete questionnaires on paper.
17. Clinically significant laboratory abnormalities.
18. History of malignancy of any organ system, treated or untreated.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
EASI value | 12 weeks
  Eczema Area and Severity Index: Each body region has potentially 100% involvement. Using the table below, give each respective body region a score of between 0 and 6 based on the percentage involvement. Precise measurements are not required.
  % involvement 0 1-9% 10 - 29% 30 - 49% 50 - 69% 70 - 89% 90 - 100% Region score 0 1 2 3 4 5 6

SECONDARY OUTCOMES:
SCORAD | 12 weeks
  Scoring Atopic Dermatitis which ranges from 0 to 103, with higher scores indicating more severe disease

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chung Wei, MD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No